CLINICAL TRIAL: NCT03388008
Title: A Pilot Randomized Controlled Trial of De Novo Belatacept-Based Immunosuppression in Lung Transplantation
Brief Title: Belatacept Pilot Study in Lung Transplantation Immunosuppression in Lung Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bela Lung Pilot
Record Dates: First submitted 2017-12-18; First posted 2018-01-02 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Lung Transplant Rejection; Antibody-mediated Rejection
Keywords: donor-specific HLA antibodies; lung transplantation
MeSH Terms: interventions — Abatacept; Tacrolimus; thymoglobulin; Mycophenolic Acid; Methylprednisolone; Methylprednisolone Hemisuccinate; Prednisone

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized to 1 of 2 arms: Belatacept-based immunosuppression or standard of care immunosuppression
Who Masked: Outcomes Assessor
Masking Description: Investigators examining lung biopsy results and blood for the development of donor-specific HLA antibodies will be blinded to study participants' treatment arm assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (Active Comparator): Tacrolimus + Mycophenolate mofetil + prednisone from day 0 through day 365
  Interventions: Drug: Tacrolimus; Drug: ATG; Drug: Mycophenolate Mofetil; Drug: Methylprednisolone; Drug: Prednisone
- Belatacept-based immunosuppression (Experimental): Belatacept + Tacrolimus + prednisone from day 0 through day 89, then Belatacept + Mycophenolate mofetil + prednisone from day 90 through day 365
  Interventions: Drug: Belatacept; Drug: ATG; Drug: Mycophenolate Mofetil; Drug: Methylprednisolone; Drug: Prednisone

INTERVENTIONS:
Drug: Belatacept — Belatacept will be dosed at 10 mg/kg of actual body weight on days 0, 7, 14, 28, 56, and 84 then at 5 mg/kg on day 112 and every 28 days through day 364 (i.e., on days 140, 168, 196, 224, 252, 280, 308, 336, and 364)
  Other Names: Nulojix
  Arms: Belatacept-based immunosuppression
Drug: Tacrolimus — Tacrolimus will be dosed enterally or sublingually within 48 hours of transplantation and the dose will be adjusted to target a trough blood level of 8-15 ng/ml
  Other Names: Prograf
  Arms: Standard of care
Drug: ATG — Anti-thymocyte globulin will be dosed intravenously at 3 mg/kg divided into 3 daily doses starting on day 0 after transplantation
  Other Names: Thymoglobulin
Drug: Mycophenolate Mofetil — Mycophenolate mofetil will be dosed at 1000 mg twice daily (or if the enteric coated formulation is used, this will be dosed at 720 mg twice daily. In the standard of care arm, mycophenolate mofetil will be initiated on day 0 after transplantation, whereas in the belatacept-based immunosuppression arm, mycophenolate mofetil will be initiated on day 90 after transplantation
  Other Names: Cellcept, Myfortic
Drug: Methylprednisolone — Methylprednisolone 500 mg will be given intravenously before perfusion of the allograft during the transplant procedure, then methylprednisolone 0.5 mg/kg will be given intravenously twice daily for 6 total doses
  Other Names: Solumedrol
Drug: Prednisone — Prednisone will be dosed at 0.5 mg/kg orally daily through day 14, then 0.2 mg/kg orally daily through day 30, then 0.1 mg/kg daily through day 180, then 5 mg daily through day 365

SUMMARY:
This is a pilot randomized controlled trial examining the feasibility of conducting a large scale randomized controlled trial of belatacept-based immunosuppression in lung transplantation. This pilot study will enroll 40 lung transplant recipients and randomize them to belatacept-based immunosuppression or standard of care. The primary endpoint of the study is the development of donor-specific HLA antibodies after transplantation. All study participants will be followed for a minimum of 12 months after transplantation.

DETAILED DESCRIPTION:
Lung transplantation is the ultimate treatment for patients with advanced lung disease. However, long-term outcomes remain disappointing and the median survival after transplantation is approximately 5.5 years. Beyond the first year after transplantation, chronic lung allograft dysfunction is the leading cause of death. The exact mechanisms that lead to chronic lung allograft dysfunction are unclear, but the development of donor-specific HLA antibodies is an independent risk factor. In fact, studies have consistently identified the development of donor-specific HLA antibodies as a significant and independent risk factor for chronic lung allograft dysfunction and mortality after transplantation.

Belatacept is a CTLA4-Ig fusion protein that binds CD80 and CD86 thereby blocking CD28 co-stimulatory signals. Belatacept has been extensively studied in kidney transplantation. In a long-term study, patients treated with Belatacept had better survival than those treated with Cyclosporine. Importantly, Belatacept-treated patients were significantly less likely to develop donor-specific HLA antibodies than Cyclosporine-treated patients. Nonetheless, Belatacept has not been formally evaluated after lung transplantation. The investigators hypothesize that Belatacept-based immunosuppression would result in a lower incidence of donor-specific HLA antibodies and that this would result in better chronic lung allograft dysfunction-free survival after transplantation. Before conducting a large scale randomized controlled trial to test this hypothesis, the investigators plan to conduct the current pilot randomized controlled trial to examine the feasibility of conducting the large scale randomized controlled trial.

The investigators plan to enroll and randomize 40 lung transplant recipients at 2 sites. All recipients will be treated with anti-thymocyte globulin for induction immunosuppression. Those randomized to standard of care immunosuppression will be treated with Tacrolimus, Mycophenolate mofetil, and prednisone. Those randomized to Belatacept-based immunosuppression will be treated with Belatacept, Tacrolimus, and prednisone for the first 89 days; on day 90, Mycophenolate mofetil will be substituted for Tacrolimus and patients will be continued on Belatacept, Mycophenolate mofetil, and prednisone for the remainder of year 1 after transplantation.

Patients in both groups will be monitored closely for episodes of acute cellular rejection, lymphocytic bronchiolitis, and antibody-mediated rejection with surveillance bronchoscopy and transbronchial lung biopsies on days 28, 84, 112, 168, 252, and 365 (± 7 days) as part of the sites' routine clinical protocols. In addition, patients will be monitored for the development of donor-specific HLA antibodies with routine blood tests on on days 10 (± 3 days), 28, 56, 84, 112, 168, 252, and 365 (± 7 days).

The primary endpoint of the study is a composite of the development of donor-specific HLA antibodies, re-transplantation, and death. Secondary endpoints include acute cellular rejection, lymphocytic bronchiolitis, antibody-mediated rejection, chronic lung allograft dysfunction, survival, cytomegalovirus infection, bacterial infection, community-acquired respiratory viral infection, chronic kidney disease stage 3, malignancy, hypertension, diabetes, and hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Provided written informed consent for study participation
* Underwent single or bilateral lung transplantation
* Negative urine pregnancy test for women of child bearing potential and willingness to use highly-effective contraception

Exclusion Criteria:

* Requiring invasive mechanical ventilation immediately before transplantation
* Requiring extracorporeal life support (ECLS) (i.e., ECMO) immediately before transplantation
* Received treatment to deplete HLA antibodies before transplantation to improve the possibility of transplantation
* Having DSA immediately before transplantation (i.e., positive virtual crossmatch)
* Listed for multi-organ transplant (e.g., heart-lung, liver-lung, kidney-lung)
* Pregnant or breast-feeding
* Active infection with Hepatitis B or C virus
* Active infection with human immunodeficiency virus (HIV)
* Chronic infection with Burkholderia cepacia complex before transplantation
* Epstein Barr Virus (EBV) seronegative status
* Participation in another interventional clinical trial
* Allograft dysfunction requiring ECMO support after transplantation
* Delayed chest closure after transplantation
* Severe coagulopathy and significant bleeding in the opinion of the PI
* Any condition that in the opinion of the site PI introduces undue risk by participating in this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramsey R Hachem, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yusen RD, Edwards LB, Kucheryavaya AY, Benden C, Dipchand AI, Goldfarb SB, Levvey BJ, Lund LH, Meiser B, Rossano JW, Stehlik J. The Registry of the International Society for Heart and Lung Transplantation: Thirty-second Official Adult Lung and Heart-Lung Transplantation Report--2015; Focus Theme: Early Graft Failure. J Heart Lung Transplant. 2015 Oct;34(10):1264-77. doi: 10.1016/j.healun.2015.08.014. Epub 2015 Sep 3. No abstract available. PMID 26454740
- [Background] Estenne M, Maurer JR, Boehler A, Egan JJ, Frost A, Hertz M, Mallory GB, Snell GI, Yousem S. Bronchiolitis obliterans syndrome 2001: an update of the diagnostic criteria. J Heart Lung Transplant. 2002 Mar;21(3):297-310. doi: 10.1016/s1053-2498(02)00398-4. No abstract available. PMID 11897517
- [Background] Verleden GM, Raghu G, Meyer KC, Glanville AR, Corris P. A new classification system for chronic lung allograft dysfunction. J Heart Lung Transplant. 2014 Feb;33(2):127-33. doi: 10.1016/j.healun.2013.10.022. Epub 2013 Oct 24. PMID 24374027
- [Background] Meyer KC, Raghu G, Verleden GM, Corris PA, Aurora P, Wilson KC, Brozek J, Glanville AR; ISHLT/ATS/ERS BOS Task Force Committee; ISHLT/ATS/ERS BOS Task Force Committee. An international ISHLT/ATS/ERS clinical practice guideline: diagnosis and management of bronchiolitis obliterans syndrome. Eur Respir J. 2014 Dec;44(6):1479-503. doi: 10.1183/09031936.00107514. Epub 2014 Oct 30. PMID 25359357
- [Background] Lama VN, Murray S, Lonigro RJ, Toews GB, Chang A, Lau C, Flint A, Chan KM, Martinez FJ. Course of FEV(1) after onset of bronchiolitis obliterans syndrome in lung transplant recipients. Am J Respir Crit Care Med. 2007 Jun 1;175(11):1192-8. doi: 10.1164/rccm.200609-1344OC. Epub 2007 Mar 8. PMID 17347496
- [Background] Finlen Copeland CA, Snyder LD, Zaas DW, Turbyfill WJ, Davis WA, Palmer SM. Survival after bronchiolitis obliterans syndrome among bilateral lung transplant recipients. Am J Respir Crit Care Med. 2010 Sep 15;182(6):784-9. doi: 10.1164/rccm.201002-0211OC. Epub 2010 May 27. PMID 20508211
- [Background] Singer JP, Singer LG. Quality of life in lung transplantation. Semin Respir Crit Care Med. 2013 Jun;34(3):421-30. doi: 10.1055/s-0033-1348470. Epub 2013 Jul 2. PMID 23821515
- [Background] Daud SA, Yusen RD, Meyers BF, Chakinala MM, Walter MJ, Aloush AA, Patterson GA, Trulock EP, Hachem RR. Impact of immediate primary lung allograft dysfunction on bronchiolitis obliterans syndrome. Am J Respir Crit Care Med. 2007 Mar 1;175(5):507-13. doi: 10.1164/rccm.200608-1079OC. Epub 2006 Dec 7. PMID 17158279
- [Background] Glanville AR, Aboyoun CL, Havryk A, Plit M, Rainer S, Malouf MA. Severity of lymphocytic bronchiolitis predicts long-term outcome after lung transplantation. Am J Respir Crit Care Med. 2008 May 1;177(9):1033-40. doi: 10.1164/rccm.200706-951OC. Epub 2008 Feb 8. PMID 18263803
- [Background] Hachem RR, Khalifah AP, Chakinala MM, Yusen RD, Aloush AA, Mohanakumar T, Patterson GA, Trulock EP, Walter MJ. The significance of a single episode of minimal acute rejection after lung transplantation. Transplantation. 2005 Nov 27;80(10):1406-13. doi: 10.1097/01.tp.0000181161.60638.fa. PMID 16340783
- [Background] Le Pavec J, Suberbielle C, Lamrani L, Feuillet S, Savale L, Dorfmuller P, Stephan F, Mussot S, Mercier O, Fadel E. De-novo donor-specific anti-HLA antibodies 30 days after lung transplantation are associated with a worse outcome. J Heart Lung Transplant. 2016 Sep;35(9):1067-77. doi: 10.1016/j.healun.2016.05.020. Epub 2016 May 31. PMID 27373824
- [Background] Tikkanen JM, Singer LG, Kim SJ, Li Y, Binnie M, Chaparro C, Chow CW, Martinu T, Azad S, Keshavjee S, Tinckam K. De Novo DQ Donor-Specific Antibodies Are Associated with Chronic Lung Allograft Dysfunction after Lung Transplantation. Am J Respir Crit Care Med. 2016 Sep 1;194(5):596-606. doi: 10.1164/rccm.201509-1857OC. PMID 26967790
- [Background] Girnita AL, McCurry KR, Iacono AT, Duquesnoy R, Corcoran TE, Awad M, Spichty KJ, Yousem SA, Burckart G, Dauber JH, Griffith BP, Zeevi A. HLA-specific antibodies are associated with high-grade and persistent-recurrent lung allograft acute rejection. J Heart Lung Transplant. 2004 Oct;23(10):1135-41. doi: 10.1016/j.healun.2003.08.030. PMID 15477106
- [Background] Girnita AL, Duquesnoy R, Yousem SA, Iacono AT, Corcoran TE, Buzoianu M, Johnson B, Spichty KJ, Dauber JH, Burckart G, Griffith BP, McCurry KR, Zeevi A. HLA-specific antibodies are risk factors for lymphocytic bronchiolitis and chronic lung allograft dysfunction. Am J Transplant. 2005 Jan;5(1):131-8. doi: 10.1111/j.1600-6143.2004.00650.x. PMID 15636621
- [Background] Bharat A, Kuo E, Steward N, Aloush A, Hachem R, Trulock EP, Patterson GA, Meyers BF, Mohanakumar T. Immunological link between primary graft dysfunction and chronic lung allograft rejection. Ann Thorac Surg. 2008 Jul;86(1):189-95; discussion 196-7. doi: 10.1016/j.athoracsur.2008.03.073. PMID 18573422
- [Background] Jaramillo A, Smith CR, Maruyama T, Zhang L, Patterson GA, Mohanakumar T. Anti-HLA class I antibody binding to airway epithelial cells induces production of fibrogenic growth factors and apoptotic cell death: a possible mechanism for bronchiolitis obliterans syndrome. Hum Immunol. 2003 May;64(5):521-9. doi: 10.1016/s0198-8859(03)00038-7. PMID 12691702
- [Background] Maruyama T, Jaramillo A, Narayanan K, Higuchi T, Mohanakumar T. Induction of obliterative airway disease by anti-HLA class I antibodies. Am J Transplant. 2005 Sep;5(9):2126-34. doi: 10.1111/j.1600-6143.2005.00999.x. PMID 16095491
- [Background] Fukami N, Ramachandran S, Saini D, Walter M, Chapman W, Patterson GA, Mohanakumar T. Antibodies to MHC class I induce autoimmunity: role in the pathogenesis of chronic rejection. J Immunol. 2009 Jan 1;182(1):309-18. doi: 10.4049/jimmunol.182.1.309. PMID 19109162
- [Background] Mohan S, Palanisamy A, Tsapepas D, Tanriover B, Crew RJ, Dube G, Ratner LE, Cohen DJ, Radhakrishnan J. Donor-specific antibodies adversely affect kidney allograft outcomes. J Am Soc Nephrol. 2012 Dec;23(12):2061-71. doi: 10.1681/ASN.2012070664. Epub 2012 Nov 15. PMID 23160511
- [Background] Vincenti F, Larsen C, Durrbach A, Wekerle T, Nashan B, Blancho G, Lang P, Grinyo J, Halloran PF, Solez K, Hagerty D, Levy E, Zhou W, Natarajan K, Charpentier B; Belatacept Study Group. Costimulation blockade with belatacept in renal transplantation. N Engl J Med. 2005 Aug 25;353(8):770-81. doi: 10.1056/NEJMoa050085. PMID 16120857
- [Background] Vincenti F, Charpentier B, Vanrenterghem Y, Rostaing L, Bresnahan B, Darji P, Massari P, Mondragon-Ramirez GA, Agarwal M, Di Russo G, Lin CS, Garg P, Larsen CP. A phase III study of belatacept-based immunosuppression regimens versus cyclosporine in renal transplant recipients (BENEFIT study). Am J Transplant. 2010 Mar;10(3):535-46. doi: 10.1111/j.1600-6143.2009.03005.x. PMID 20415897
- [Background] Vincenti F, Larsen CP, Alberu J, Bresnahan B, Garcia VD, Kothari J, Lang P, Urrea EM, Massari P, Mondragon-Ramirez G, Reyes-Acevedo R, Rice K, Rostaing L, Steinberg S, Xing J, Agarwal M, Harler MB, Charpentier B. Three-year outcomes from BENEFIT, a randomized, active-controlled, parallel-group study in adult kidney transplant recipients. Am J Transplant. 2012 Jan;12(1):210-7. doi: 10.1111/j.1600-6143.2011.03785.x. Epub 2011 Oct 12. PMID 21992533
- [Background] Streitz M, Miloud T, Kapinsky M, Reed MR, Magari R, Geissler EK, Hutchinson JA, Vogt K, Schlickeiser S, Kverneland AH, Meisel C, Volk HD, Sawitzki B. Standardization of whole blood immune phenotype monitoring for clinical trials: panels and methods from the ONE study. Transplant Res. 2013 Oct 25;2(1):17. doi: 10.1186/2047-1440-2-17. PMID 24160259
- [Derived] Huang HJ, Schechtman K, Askar M, Bernadt C, Mitter B, Dore P, Goodarzi A, Yau S, Youssef JG, Witt CA, Byers DE, Vazquez-Guillamet R, Halverson L, Nava R, Puri V, Kreisel D, Gelman AE, Hachem RR. A Pilot Randomized Controlled Trial of De Novo Belatacept-based Immunosuppression After Lung Transplantation. Transplantation. 2024 Mar 1;108(3):777-786. doi: 10.1097/TP.0000000000004841. Epub 2024 Feb 20. PMID 37899481

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 2 centers (Washington University in St. Louis and Houston Methodist Hospital) between 12/2019 and 5/2021.
Period: Overall Study
Arm/Group | Standard of Care | Belatacept-based Immunosuppression
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Belatacept-based Immunosuppression | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (11.8) | 57.8 (7.5) | 58.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27
Diagnosis [Count of Participants; unit: Participants]
  Interstitial Lung Disease | 8 | 7 | 15
  COPD | 0 | 4 | 4
  Pulmonary Arterial Hypertension | 2 | 0 | 2
  Other | 4 | 2 | 6
Operation [Count of Participants; unit: Participants]
  Bilateral lung transplant | 11 | 12 | 23
  Single lung transplant | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Donor-specific HLA Antibodies, Re-transplantation, or Death
Description: The Outcome Measure is a composite primary endpoint of the development of donor-specific HLA antibodies, re-transplantation, or death. Testing for donor-specifc HLA antibodies was performed at study-specified time points using the single antigen bead assay at the study core lab. Donor-specific HLA antibodies were defined as reactivity with a mean fluorescence intensity (MFI) ≥ 2,000.
Time Frame: 365 days
Measure: Number; unit: participants
Arm/Group | Standard of Care | Belatacept-based Immunosuppression
Number analyzed (Participants) | 14 | 13
participants
  Death | 0 | 5
  Donor-specific HLA antibodies | 3 | 3
  Re-transplantation | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 14 months after randomization. However, not all participants have completed 14 months of follow-up at this time.
Arm/Group | Standard of Care | Belatacept-based Immunosuppression
All-Cause Mortality (participants affected / at risk) | 0/14 | 5/13
Serious Adverse Events (participants affected / at risk) | 10/14 | 10/13
Other Adverse Events (participants affected / at risk) | 12/14 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=14) | Belatacept-based Immunosuppression (N=13)
Venous Thromboembolism (Vascular disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (12)
COVID-19 infection (Infections and infestations) | 3 (3) | 2 (2)
Surgical site infection (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Acute rejection (Immune system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Limb ischemia (Vascular disorders) | 1 (1) | 0 (0)
Nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Parainfluenza virus infection (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Post-transplant lymphoproliferative disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Multiple fractures (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=14) | Belatacept-based Immunosuppression (N=13)
Ischemic mucosal airway injury (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Pulmonary nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchomalacia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diaphragmatic dysfunction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Anastomotic air leak (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary eosinophilia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Positive bronchoscopy culture (Infections and infestations) | 9 (31) | 8 (13)
Upper respiratory infection (Infections and infestations) | 1 (1) | 2 (4)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Mucocutaneous HSV (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Acute cellular rejection (Immune system disorders) | 7 (7) | 3 (4)
Hypogammaglobulinemia (Immune system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 6 (6)
Hypotension (Vascular disorders) | 3 (3) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Hypovolemia (Vascular disorders) | 1 (1) | 0 (0)
Aortic root dilation (Vascular disorders) | 1 (1) | 0 (0)
Cardiac dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Orthostasis (Vascular disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric distention (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
GERD (Gastrointestinal disorders) | 0 (0) | 1 (1)
Electrolyte abnormality (Renal and urinary disorders) | 7 (7) | 5 (6)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 8 (8) | 9 (10)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Delirium (Nervous system disorders) | 2 (2) | 3 (3)
Gait abnormality (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Generalized weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Calf pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Calcific panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Edema (Vascular disorders) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Hoarseness (General disorders) | 1 (1) | 0 (0)
Vocal cord dysfunction (General disorders) | 2 (2) | 0 (0)
Dysphonia (General disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Endocrine disorders) | 2 (2) | 1 (1)
Hypercholesterolemia (Endocrine disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Wound dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT03388008/Prot_SAP_000.pdf